CLINICAL TRIAL: NCT06900231
Title: Knowledge, Attitudes, and Beliefs About Musculoskeletal Pain Among Primary Care Health Professionals in Different Autonomous Communities of Spain: A Cross-Sectional Study
Brief Title: Knowledge, Attitudes, and Beliefs About Musculoskeletal Pain Among Primary Care Health Professionals in Spain.
Acronym: CACDAPES
Status: Not yet recruiting | Type: Observational
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Francesc Valenzuela Pascual, Associated professor, Universitat de Lleida
Other Study IDs: CACDAPES-ULleida
Record Dates: First submitted 2025-03-14; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Fear Avoidance
Keywords: Pain Management; Primary Health Care; Musculoskeletal Pain; Health Professionals; Fear-Avoidance; Pain Neurophysiology Knowledge
MeSH Terms: conditions — Agnosia; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Pain is a multifactorial experience where psychological and emotional factors influence the transition from acute to chronic pain, prognosis, and the adoption of inappropriate self-management strategies. In addition to psychological and emotional factors, healthcare professionals can contribute to the development of chronic disabilities in their patients by promoting hypervigilance and restricting normal activities, potentially reinforcing or altering patients' perceptions, leading to limited mobility. Existing scientific literature suggests that patients with chronic pain often feel they do not receive sufficient information from healthcare professionals that could help them better understand and manage pain, thereby improving their quality of life.

Objectives:

1. To assess the current knowledge of pain neurophysiology among primary care professionals (medicine, physiotherapy, nursing, nutrition, and psychology) in Spain.
2. To evaluate attitudes and beliefs about chronic low back pain among primary care professionals (medicine, physiotherapy, nursing, nutrition, and psychology) in Spain.
3. To examine fear-avoidance beliefs related to pain among primary care professionals (medicine, physiotherapy, nursing, nutrition, and psychology) in Spain.

Methodology: A cross-sectional descriptive study will be conducted to collect information from primary care health professionals (medicine, physiotherapy, psychology, nutrition, and nursing) in Spain, focusing on their current knowledge, attitudes, and beliefs about musculoskeletal pain.

Applicability: This study will provide valuable insights into the current state of knowledge, attitudes, and beliefs about musculoskeletal pain among primary care health professionals in Spain. The findings will guide future educational interventions and policy recommendations to improve the management of musculoskeletal pain in primary care settings in Spain.

Relevance: Scientifically, this will be the first study to evaluate the knowledge of primary care health professionals in Spain regarding pain neurophysiology, attitudes and beliefs about chronic low back pain, and fear-avoidance attitudes.

DETAILED DESCRIPTION:
Background: Pain is a multifactorial experience where psychological and emotional factors influence the transition from acute to chronic pain, prognosis, and the adoption of inappropriate self-management strategies. In addition to psychological and emotional factors, healthcare professionals can contribute to the development of chronic disabilities in their patients by promoting hypervigilance and restricting normal activities, potentially reinforcing or altering patients' perceptions, leading to limited mobility. Existing scientific literature suggests that patients with chronic pain often feel they do not receive sufficient information from healthcare professionals that could help them better understand and manage pain, thereby improving their quality of life.

Objectives:

1. To assess the current knowledge of pain neurophysiology among primary care professionals (medicine, physiotherapy, nursing, nutrition, and psychology) in Spain.
2. To evaluate attitudes and beliefs about chronic low back pain among primary care professionals (medicine, physiotherapy, nursing, nutrition, and psychology) in Spain.
3. To examine fear-avoidance beliefs related to pain among primary care professionals (medicine, physiotherapy, nursing, nutrition, and psychology) in Spain.

Methodology: A cross-sectional descriptive study will be conducted to collect information from primary care health professionals (medicine, physiotherapy, psychology, nutrition, and nursing) in Spain, focusing on their current knowledge, attitudes, and beliefs about musculoskeletal pain.

Applicability: This study will provide valuable insights into the current state of knowledge, attitudes, and beliefs about musculoskeletal pain among primary care health professionals in Spain. The findings will guide future educational interventions and policy recommendations to improve the management of musculoskeletal pain in primary care settings in Spain.

Relevance: Scientifically, this will be the first study to evaluate the knowledge of primary care health professionals in Spain regarding pain neurophysiology, attitudes and beliefs about chronic low back pain, and fear-avoidance attitudes.

ELIGIBILITY:
Inclusion Criteria:

* Graduates in medicine or residents specializing in family and community medicine.

Graduates in physiotherapy. Graduates in nursing or residents specializing in family and community nursing. Graduates in psychology. Graduates in nutrition.

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Professionals in medicine, physiotherapy, nursing, psychology, and nutrition working in Primary Care Centers in Spain
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Pain Neurophysiology Knowledge Questionnaire | One-time assessment at enrollment
  The questionnaire consists of 19 questions that require true, false, or undecided answers, with a maximum score of 19 points. Higher scores mean better knowledge.

SECONDARY OUTCOMES:
HC-PAIRS | One-time assessment at enrollment
  The questionnaire consists of 15 statements on a 7-point Likert scale (1 = completely disagree, 4 = neither agree nor disagree, and 7 = completely agree), with a maximum score of 105 points. Higher scores indicate a greater degree of beliefs about the relationship between chronic pain, functional limitation, and disability.
Fear-Avoidance believes | One-time assessment at enrollment
  The questionnaire is divided into two subscales, FABQ-Physical Activity (questions 1-5) and FABQ-Work (questions 6-16), and consists of a total of 16 statements that require responses on a 6-point Likert scale (0 = completely disagree and 6 = completely agree), with a maximum score of 96 points. Higher scores indicate a greater degree of fear-avoidance beliefs.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat de Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: Undecided